CLINICAL TRIAL: NCT03797794
Title: The Influence of Pulsating Electrostatic Field (PESF) on Oxygen Saturation, Quality of Life and Exercise Capacity of COPD Patients, a Single Center, Double Blind, Placebo Controlled Study.
Brief Title: Influence of PESF on Oxygen Saturation, Quality of Life and Exercise Capacity in COPD
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Logistical problems at study site
Sponsor: University Medical Center Groningen (Other)
Collaborators: Tjongerschans hospital (Unknown)
Responsible Party: Principal Investigator, Huib A.M. Kerstjens, Head of the department Pulmonary diseases and Tuberculosis, University Medical Center Groningen
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: PESF and COPD
Record Dates: First submitted 2019-01-07; First posted 2019-01-09 (Actual); Last update posted 2024-01-19 (Actual); Status verified 2024-01

CONDITIONS: COPD
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Intervention Model Description: prospective, randomized, dubbel blind, placebo-controlled parallel study
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PESF-treatment (Experimental): The group undergoing the pulsating electrostatic field intervention
  Interventions: Device: Pulsating Electrostatic Field
- Placebo-treatment (Sham Comparator): The group undergoing the SHAM Pulsating Electrostatic Field
  Interventions: Device: SHAM Pulsating Electrostatic Field

INTERVENTIONS:
Device: Pulsating Electrostatic Field — A pulsating electrostatic field is generated by the New Health 9000 (Akern). During the session the patients sits on a chair which contains the apparatus for 30 minutes.
  Arms: PESF-treatment
Device: SHAM Pulsating Electrostatic Field — The same apparatus which produces the pulsating electrostatic field contains a 'sham-inlet'. This inlet will be used as placebo.
  Arms: Placebo-treatment

SUMMARY:
The effect of PESF (Pulsating Electrostatic Field) on the oxygen saturation, quality of life and the exercise capacity will be studied in a randomized, dubbel blind, placebo-controlled parallel design with 32 COPD patients GOLD III and IV with a oxygen saturation below or equal to 90%.

The patients will be treated with three 30-minute PESF- or placebo-sessions distributed over 5 days.

Directly before the first session, oxygen saturation, quality of life (CCQuestionnaire), exercise capacity (6-MWT and grip strength) and phase angle (BIA) will be measured and compared to the results directly after the third session. Oxygen saturation is also monitored during 24 hours after each session.

ELIGIBILITY:
Inclusion Criteria:

* COPD patients, post-bronchodilator FEV1/FVC <70% and FEV1 <50% predicted
* oxygen saturation without suppletion <=90% (home use of oxygen suppletion is allowed, but will be stopped during PESF-treatment)
* Stable medication (no foreseeable need to change therapy)
* Able to understand the purpose and method of research after adequate information and the ability to decide on participation
* Signed informed consent

Exclusion Criteria:

* Known malignant condition with limited life expectancy
* Carrier of electrical equipment (pacemaker, ICD etc)
* COPD exacerbation in the last 3 weeks
* Woman who are pregnant or of childbearing age without effective contraception
* Manifest acute infection
* Patients with manifest decompensatio cordis
* Rehabilitation/reactivation program within 2 months before or during the study

Ages: 40 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Improvement of oxygen saturation | 5 days
  Difference in oxygen saturation before first vs after last session

SECONDARY OUTCOMES:
Improvement of quality of life | 5 days
  Difference in CCQ score before first vs after last session
Improvement of exercise capacity | 5 days
  Difference in 6-MWT outcome before first vs after last session
Improvement of phase angle | 5 days
  Difference in oxygen saturation before first vs after last session

CONTACTS AND LOCATIONS:
Locations (1):
- Tjongerschans, Heerenveen, Provincie Friesland, Netherlands